CLINICAL TRIAL: NCT00154011
Title: Characterization of Vascular Effects of Rosiglitazone.
Brief Title: Investigation of Vascular Relaxing Effects of the Antidiabetic Rosiglitazone.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Technische Universität Dresden (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IKPD 01-05
Record Dates: First submitted 2005-09-08; First posted 2005-09-12 (Estimated); Last update posted 2006-09-12 (Estimated); Status verified 2006-09

CONDITIONS: Healthy Subjects
Keywords: vascular reactivity, venodilation
MeSH Terms: interventions — Rosiglitazone; Pharmaceutical Preparations

INTERVENTIONS:
Drug: rosiglitazone (drug)

SUMMARY:
The study is designed to test the hypothesis in healthy subjects that the oral antidiabetic drug rosiglitazone provides additional vascular relaxing or modulating effects in addition to its blood glucose level reducing ability.

DETAILED DESCRIPTION:
The aim of the study is to investigate the effect of oral rosiglitazone therapy on the vascular responsiveness of different vasoactive compounds (angiotensin II, insulin, histamine and glyceroltrinitrate) in healthy subjects. Rosiglitazone will be given orally (4 weeks 4mg/d, titrated to 8 mg/d for another 4 weeks) as treatment. Every subject will receive intravenous stimulation with angiotensin II, histamine, insulin and glyceroltrinitrate before and after an 8 weeks treatment interval with rosiglitazone.

ELIGIBILITY:
Inclusion Criteria:

* Male
* Healthy
* 18 - 40 years old
* Non-smoker
* No additional medication

Exclusion Criteria:

* Any relevant disease
* Smokers
* Elevated liver enzymes
* Body weight different from Broca norm > 20%
* Allergies

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24
Dates: Start 2005-09; Study Completion 2006-06

PRIMARY OUTCOMES:
Vascular reactivity after 8 weeks treatment.

SECONDARY OUTCOMES:
Changes in angiotensin peptide metabolism.

CONTACTS AND LOCATIONS:
Overall Officials: Wilhelm Kirch, MD, Study Chair — Institute of Clinical Pharmacology
Locations (1):
- Institute of Clinical Pharmacology, Dresden, Germany